CLINICAL TRIAL: NCT07277166
Title: The Effect of Mobile Robot Assisted Gait Training on Gait Performance in Chronic Patients With Impaired Gait Function After Burn Injury : Pilot Study
Brief Title: The Effect of Mobile Robot Assisted Gait Training on Gait Performance in Chronic Patients With Impaired Gait Function After Burn Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hangang Sacred Heart Hospital (Other)
Responsible Party: Principal Investigator, So Young Joo, Principal Investigator, Department of rehabilitation medicine of Hangang Sacred heart hospial, Hangang Sacred Heart Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HangangSHH-22
Record Dates: First submitted 2025-11-25; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Burns; Gait Dysfunction; Robot Training
Keywords: BURNS, Gait dysfunction, Wearable robot, Robot training
MeSH Terms: conditions — Burns

STUDY DESIGN:
Intervention Model Description: The wearable robot (WIRobotics Inc) is a wearable robot designed to provide assistive torque and resistive torque for hip movement. It is worn around the waist and thighs and weight approximately 1.6 kg. The main body and actuation parts are not located at the hip joints and back to avoid restricting body movements and to facilitate movement even in cramped spaces.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Wearable robot training (Experimental): The wearable robot (WIRobotics Inc) is a wearable robot designed to provide assistive torque and resistive torque for hip movement. It is worn around the waist and thighs and weight approximately 1.6 kg. The main body and actuation parts are not located at the hip joints and back to avoid restricting body movements and to facilitate movement even in cramped spaces. Physiotherapy was performed on a one to one basis by qualified physiotherapists for 1 hour per day, 5 days a week Monday through Friday, for 12 weeks.
  Interventions: Other: wearable robot training

INTERVENTIONS:
Other: wearable robot training — The wearable robot (WIRobotics Inc) is a wearable robot designed to provide assistive torque and resistive torque for hip movement. It is worn around the waist and thighs and weight approximately 1.6 kg. The main body and actuation parts are not located at the hip joints and back to avoid restricting body movements and to facilitate movement even in cramped spaces. Physiotherapy was performed on a one to one basis by qualified physiotherapists for 1 hour per day, 5 days a week Monday through Friday, for 12 weeks.

SUMMARY:
This study aims to examine the clinical effectiveness of gait training using wearable robots in patients with impaired gait function after burn injury. The participants were chronic patients who underwent split-thickness skin grafting or burns of more than 50% of the lower extremities and still had impaired gait dysfunction 6 months later. Eligible participants were aged over 18 years and had a Functional Ambulation Category (FAC) score of 3 or higher. Physiotherapy was performed on a one to one basis by qualified physiotherapists for 1 hour per day, 5 days a week Monday through Friday, for 12 weeks. Assessments were carried out before and immediately after the 12-week training period. Physical ability were assessed using the functional ambulatory category(FAC) scale, the 6-Minute Walk Test (6MWT), and the visual analogue scale (VAS). Spatiotemporal gait parameters-including gait speed, cadence, and step length-and sagittal joint kinematic parameters for the hip, knee, and ankle during stance and swing phases were measured during gait analysis. Pulmonary function test such as forced vital capacity (FVC), 1-s forced expiratory volume (FEV1), and carbon monoxide (DLco). The highest maximal expiratory pressure (MEP) and maximal inspiratory pressure (MIP) value were evaluated.

DETAILED DESCRIPTION:
Regaining a mobility level post-surgery that comes close to the patient's previous mobility as a baseline is the goal. It is commonly accepted that conventional physiotherapy after burn injury has a positive impact on muscle strength, range of motion, pain or gait performance which all impact patient mobility. Wearable robots that assist walking centered on the hip joint of the lower extremities are appearing. This wearable robot is a positive effect in terms of increased energy efficiency and posture during walking. This study aims to examine the clinical effectiveness of gait training using wearable robots in patients with impaired gait function after burn injury. The participants were chronic patients who underwent split-thickness skin grafting or burns of more than 50%of the lower extremities and still had impaired gait dysfunction 6 months later. Eligible participants were aged over 18 years and had a Functional Ambulation Category (FAC) score of 3 or higher. This study excluded patients with fourth-degree burns (involving muscles, tendons, and bone injuries), severe communication disorders because of intellectual impairment and psychological problems. The specific exclusion criteria were as follows. Patients with body types that prevent them form wearing the robot, such as a height of 4.59 feet (140cm) or 5.91 feet (185cm) or more, or severe obesity with a BMI of 35 or more. Patients with heart and circulatory conditions that may affect gait training. Patients at a high risk of falling during gait training, owing to severe dizziness and having experienced a fall within the preceeding 2 month.Physiotherapy was performed on a one to one basis by qualified physiotherapists for 1 hour per day, 5 days a week Monday through Friday, for 12 weeks. Assessments were carried out before and immediately after the 12-week training period. Physical ability were assessed using the functional ambulatory category(FAC) scale, the 6-Minute Walk Test (6MWT), and the visual analogue scale (VAS). Spatiotemporal gait parameters-including gait speed, cadence, and step length-and sagittal joint kinematic parameters for the hip, knee, and ankle during stance and swing phases were measured during gait analysis. Pulmonary function test such as forced vital capacity (FVC), 1-s forced expiratory volume (FEV1), and carbon monoxide (DLco). The highest maximal expiratory pressure (MEP) and maximal inspiratory pressure (MIP) value were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* chronic patients who underwent split-thickness skin grafting or burns of more than 50% of the lower extremities and still had impaired gait dysfunction 6 months later. -aged over 18 years
* had a Functional Ambulation Category (FAC) score of 3 or higher

Exclusion Criteria:

* fourth-degree burns (involving muscles, tendons, and bone injuries)
* severe communication disorders because of intellectual impairment and psychological problems
* Patients with body types that prevent them form wearing the robot, such as a height of 4.59 feet (140cm) or 5.91 feet (185cm) or more, or severe obesity with a BMI of 35 or more.
* Patients with heart and circulatory conditions that may affect gait training.
* Patients at a high risk of falling during gait training, owing to severe dizziness and having experienced a fall within the preceeding 2 month.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-05-13 (Actual); Primary Completion 2026-11-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
functional ambulatory category | 12 weeks
  Participants were rated on a six-point scale based on the level of physical assistance required for walking, regardless of whether an assistive device was used.

SECONDARY OUTCOMES:
6-Minute Walk Test (6MWT) | 12weeks
  conducted according to standardized guidelines, on a 20-meter walking course. Patients were instructed to walk as far as possible in 6 min.
visual analogue scale (VAS) | 12 weeks
  rate the degree of subjective pain during gait movement (0 points : when no pain was noted, and 10 points : when unbearable pain was noted).
sagittal joint kinematic parameters for the hip, knee, and ankle during stance and swing phases | 12 weeks
  the total range of motion of hip, knee, and ankle during one gait cycle

CONTACTS AND LOCATIONS:
Locations (1):
- Hangang sacred heart hodpital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
The datasets used and/or analysed during the current study are available from the corresponding author on reasonable request.

REFERENCES:
- [Result] Shin JH, Byeon N, Yu H, Lee D, Lee HJ, Lee WH. Effect of wearable robot Bot Fit's hip joint-centered assist torque and voice coach on walking. BMC Musculoskelet Disord. 2024 Dec 23;25(1):1063. doi: 10.1186/s12891-024-08181-8. PMID 39716173
- [Result] Cho E, Hwang S, Heo SJ, Lim B, Lee J, Lee Y. Feasibility and Effects of a Gait Assistance and Gait Resistance Training Program Using a Walking-Assist Wearable Robot for Community-Dwelling Older Adults: Single-Group, Pre-, and Posttest Study. JMIR Mhealth Uhealth. 2025 May 26;13:e58142. doi: 10.2196/58142. PMID 40418849